CLINICAL TRIAL: NCT06917274
Title: Effects of Pre-Exercise Banana Consumption on Glycemic Control in Individuals With Type 1 Diabetes
Brief Title: The Banana Exercise Type 1 Diabetes Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-9-25
Record Dates: First submitted 2025-03-20; First posted 2025-04-08 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Type 1 Diabetes
Keywords: nutrition; CGM; blood glucose; exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- No banana (Active Comparator): No banana consumed prior exercise
  Interventions: Other: No banana
- banana (Active Comparator): Banana consumed 20 minutes prior exercise
  Interventions: Dietary Supplement: Banana

INTERVENTIONS:
Dietary Supplement: Banana — A banana is consumed pre-exercise in order to prevent hypoglycemia
  Arms: banana
Other: No banana — No banana is consumed pre-exercise
  Arms: No banana

SUMMARY:
Former and current KADET athletes participate in two controlled training sessions: one with a banana 20 minutes pre-exercise and one without. Tandem Data recorded includes sensor glucose, training details, insulin dosing, and meal intake. Continuous glucose monitoring (CGM) data is assessed. Endpoints include differences in glucose levels, hypoglycemia events (SG <3.9 mmol/L), and Time in Range during training

DETAILED DESCRIPTION:
Participants:

Former and current KADET athletes invited via a Facebook group. Previous participants in study projects who have expressed interest in being contacted for future studies.

Protocol:

Participants provide written consent for data collection and use.

Each participant completes two training sessions under controlled conditions, including:

Same training time Standardized pre-training meal timing and insulin corrections Similar intensity and environmental factors If pre-training hypoglycemia occurs, training is rescheduled or corrected with glucose tablets, which are documented.

Study Conditions:

Session 1: Participant eats a banana 20 minutes before training. Session 2: No pre-training food intake.

Tandem Control IQ users (insulin pump) take a microbolus (0.05 IE) before banana intake.

Recorded Data by participant:

Training start and end times Sensor glucose (SG) at start and end of training Training type and intensity (Borg scale, heart rate monitoring) Last insulin dose (meal and correction) Last meal details (content and timing) Banana documentation (photo, weight with peel, ripeness level)

CGM data are also assessed.

Endpoints:

Differences in GCG glucose level Time to hypoglycemia and number of hypoglycemia events (SG <3.9 mmol/L) on banana vs. non-banana days.

Percentage of Time in Range during training. Additional data is reported as available.

ELIGIBILITY:
Inclusion Criteria:

* type 1 diabetes

Exclusion Criteria:

* cardiovascular comorbidity
* neuropathy

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
CGM glucose | approximately 60 minute monitoring period during exercise
  CGM glucose Time in Range between 3.9 and 10 mmol/l

SECONDARY OUTCOMES:
Time to hypoglycemia | approximately 30 to 30 minutes
  minutes to hypoglycemia after exercise has begun
Borg scale | Borg scale is assessed approximately 15 minutes after exercise
  Level of excaution evaluated on Borg scale from 6-20

IPD SHARING:
Plan to Share IPD: No